CLINICAL TRIAL: NCT04358250
Title: Tissue Sparing Surgery in Total Hip Arthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: I.R.C.C.S Ospedale Galeazzi-Sant'Ambrogio (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TSSINTHA2016
Record Dates: First submitted 2018-01-18; First posted 2020-04-24 (Actual); Last update posted 2020-04-24 (Actual); Status verified 2020-04

CONDITIONS: Total Hip Arthroplasty; Hip Arthrosis
Keywords: tissue sparing surgery
MeSH Terms: conditions — Osteoarthritis, Hip

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- direct superior approach (Experimental): Direct superior approach 25 patients
  Interventions: Procedure: Direct Superior Approach
- posterolateral approach (Active Comparator): posterolateral approach 25 patients
  Interventions: Procedure: posterolateral approach

INTERVENTIONS:
Procedure: Direct Superior Approach — GROUP II :Patients positioned in lateral decubitus.landmark for incision is the apex of the greater trochanter,and skin, subcutaneous tissue except fascia are incised accordingly. Fibers of gluteus will be separated and not incised.posterior capsulotomy is performed,;femur is dislocated and neck osteotomy carried out, followed by preparation of femoral canal with progressive broach. Acetabulum is prepared with burs of increasing diameter, and acetabular cup is impacted. A polyethylene insert and a femoral rasp are subsequently introduced.All remaining definitive implants can be positioned.
  Other Names: DSA
  Arms: direct superior approach
Procedure: posterolateral approach — GROUP I:patients are positioned in lateral decubitus.Landmark for incision is the apex of the greater trochanter.posterior capsulotomy is performed, femur is dislocated and neck osteotomy carried out, followed by preparation of femoral canal with progressive broach.Acetabulum is prepared with burs of increasing diameter,and acetabular cup is then impacted.All definitive implants can be positioned.
  Arms: posterolateral approach

SUMMARY:
Rationale of the study is to evaluate through a prospective randomized controlled study if a modified direct superior posterolateral approach (sperimental approach) to the hip articulation which entirely spares i.e. avoids the sacrifice of the fascia lata might elicit a better outcome in terms of gait, balance, strengths recovery, clinical performance, patient reported outcome measurement (Short Form-12(SF-12); Hip disability and Osteoarthritis Outcome Score (HOOS)) and overall recovery time in patients undergoing TotalHipArthroplasty with the aid of dedicated, modified instrumentation in order to properly access this modified route.

The investigators expect an improvement on selected gait analysis parameters in sperimental approach in order of 2% of range of motion (ROM) recorded 1 month after surgery. Based on this assumption sample size calculation will be conducted.

DETAILED DESCRIPTION:
Rationale of the study is to evaluate through a prospective randomized controlled study if a modified direct superior approach (experimental approach) to the hip articulation which entirely spares i.e. avoids the sacrifice of the fascia lata (posterolateral approach) might elicit a better outcome in terms of gait, balance,strenghts recovery, clinical performance, patient reported outcome measurements and overall recovery time in patients undergoing TotalHipArthroplasty with the aid of dedicated, modified instrumentation in order to properly access this modified route.Two patients groups will randomly be allocated in one of the two group with a computer generated 1:1 randomization table.Total number of subjects participating in the study:50.

ELIGIBILITY:
Inclusion Criteria:- Patients affected by:

* Non-inflammatory degenerative joint disease, including osteoarthritis
* Patients in the age from 60 to 85 included
* Consenting to actively participate in the study and in the rehabilitation follow up program as foreseen by the study
* 18 ≤ Body Mass Index (BMI) ≥ 30 kg/m2
* patient without contralateral THA

Exclusion Criteria:-Revision procedures where other treatments or devices have failed

* Active infection or suspected latent infection in or about the hip joint
* Bone stock that is inadequate for support or fixation of the prosthesis
* skeletal immaturity
* any mental or neuromuscular disorder that would create an unacceptable risk of prosthesis instability, prosthesis fixation failure or complication in post-operative care
* Obesity (BMI ≥30kg/m2)

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2017-04-26 (Actual); Primary Completion 2017-10-25 (Actual); Study Completion 2018-11-30 (Actual)

PRIMARY OUTCOMES:
evaluate spatiotemporal variables in meters among two different access routes, one a traditional posterolateral mini approach and the other a modified posterolateral superior approach fascia lata sparing | Change from Baseline spatiotemporal variables in meters at 3 months
  spatiotemporal variables: step length (meters), stride length (meters).
evaluate spatiotemporal variables in percentage among two different access routes, one a traditional posterolateral mini approach and the other a modified posterolateral superior approach fascia lata sparing | Change from Baseline spatiotemporal variables in percentage at 3 months
  Spatiotemporal variables: stance phase (percentage), swing phase (percentage)
evaluate kinematic parameters in degrees among two different access routes, one a traditional posterolateral mini approach and the other a modified posterolateral superior approach fascia lata sparing | Change from Baseline Kinematic parameters in degrees at 3 months
  Kinematic parameters (in degrees): hip flexion-extension ROM, hip abduction-adduction ROM, Hip rotation ROM, Hip Obliquity ROM.

SECONDARY OUTCOMES:
evaluation of instability with BEStest | Change from Baseline BESTest at 3 months
  BESTest (Balance Evaluation System Test) that evaluate the risk of fall . Each patient will be asked to wear a belt and two gloves containing the magnetic sensors and to follow the OAK device instruction.The portable device detects, on real time, the position and the orientation of each sensor. It yields a point-score from 0 to 24 and it has been shown that the relative optimal cut-off point was a 16 point-score out of 24: a point score between 17 and 24 classifies a subject as low risk who would otherwise be classified as being at medium/high risk (the duration will be approximately 10 minutes)

CONTACTS AND LOCATIONS:
Overall Officials: Michele Ulivi, Principal Investigator — IRCCS Istituto Ortopedico GaleazziMilano
Locations (2):
- Italy (2):
  - IRCCS Istituto Ortopedico Galeazzi, Milan
  - Istituto Ortopedico Galeazzi, Milan

REFERENCES:
- [Derived] Ulivi M, Orlandini L, Vitale JA, Meroni V, Prandoni L, Mangiavini L, Rossi N, Peretti GM. Direct superior approach versus posterolateral approach in total hip arthroplasty: a randomized controlled trial on early outcomes on gait, risk of fall, clinical and self-reported measurements. Acta Orthop. 2021 Jun;92(3):274-279. doi: 10.1080/17453674.2020.1865633. Epub 2021 Jan 7. PMID 33410360